CLINICAL TRIAL: NCT03393416
Title: A Single Center, Phase I Clinical Study to Evaluate the Safety of MASCT-I Combined With PD1 Antibody in Vivo for the Advanced Soild Tumor Including Gastric Cancer，Triple-negative Breast Cancer and Ovarian Cancer
Brief Title: A Phase I Clinical Study for Evaluating the Safety of MASCT-I in Advanced Soild Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HRYZ Biotech Co. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MASCT-I-1003
Record Dates: First submitted 2017-12-27; First posted 2018-01-08 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Advanced Gastric Cancer
Keywords: MASCT-I
MeSH Terms: interventions — spartalizumab; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MASCT-I or MASCT-I +PD1 antibody (Experimental): This study is divided into three stages:
  The first, second stage is the stage of the dose climbing, and the third stage is the dose expansion stage. The first stage is MASCT-I, using 3+3 design. The second stage is divided into two groups: MASCT-I+PD1 antibody in low dose group and MASCT-I+PD1 antibody in high dose group, using 3+3 design. The third stage is the dose expansion stage , 10 patients in the low or high dose group were treated with the corresponding dose group.
  Interventions: Biological: MASCT-I; Drug: PD1 antibody

INTERVENTIONS:
Biological: MASCT-I — The final products of MASCT-I(Multiple-antigen specific cell therapy) technology are dendritic cells (DC) and effector T cells.Treatment with MASCT-I alone, conducted until disease progression, intolerance or end of study.
Drug: PD1 antibody — Drug: PD1 antibody
  1mg/kg or 3mg/kg. Administration is conducted in Day1 and Day15. Conducted until disease progression, intolerance or end of study.
  Other Names: SHR-1210

SUMMARY:
This study evaluate the safety and tolerance of MASCT-I(multiple-antigen specific cell therapy) combined with PD1 antibody in patients with advanced gastric cancer who failed in first-line chemotherapy. The study is divided into three stages: the first, second stage is the stage of the dose climbing, and the third stage is the dose expansion stage. The patients would be treated with MASCT-I single drug therapy, MASCT-I+ low dose PD1 antibody therapy, and MASCT-I+ high dose PD1 antibody therapy.

DETAILED DESCRIPTION:
The multiple-antigen specific cell therapy which was developed by Hengrui Yuanzheng is optimized continuously and has been upgraded from the first-generation MASCT technology to MASCT-I. MASCT-I is to add PD1 antibody in vitro cell culture process of MASCT technology to block PD1 receptor on immunocytes, relieving the brake at immunocytes' reinfusion and interaction with tumor cells for enhancing the effectiveness of immunocytes killing tumor cells.

This is a phase I study to evaluate the safety and tolerance of MASCT-I combined with PD1 antibody in patients with advanced gastric cancer who failed in first-line chemotherapy.

About 19-28 cases patients with advanced gastric cancer are to be recruited.

This study is divided into three stages:

The first, second stage is the stage of the dose climbing, and the third stage is the dose expansion stage. The first stage is MASCT-I, using 3+3 design, if the DLT≥33.3% from the mononuclear cell collection to 14 days after the first MASCT-I infusion of T cells,the experiment will be end. If the DLT<33.3%, enter the second stage. The second stage is divided into two groups: MASCT-I+PD1 antibody in low dose group and MASCT-I+PD1 antibody in high dose group, using 3+3 design, if all patients in low dose group, the DLT≥33.3% from the mononuclear cell collection to 14 days after the first MASCT-I infusion of T cells, the experiment will be end. If DLT<33.3% began high dose group. If all the patients in the high dose group, DLT ≥33.3%, the corresponding high dose group treatment will be terminated, entered the third stage, the dose of expansion, only by low dose treatment group of 10 patients of reentry. If all the patients in the high dose group, DLT<33.3%, entered the third stage. Only 10 patients in the high dose group were treated with the corresponding high-dose group.

ELIGIBILITY:
Inclusion Criteria:

* The age is 18-70 years old.
* The written informed consent of the patient / legal representative is obtained before any program related implementation.
* Metastatic or non resectable, locally advanced gastric or gastroesophageal adenocarcinoma, confirmed by histology or cytology.
* The development of objective imaging after first-line chemotherapy (RECIST1.1);
* There were measurable lesions (according to RECIST1.1);
* Can provide tumor tissue specimens;
* PDL1 positive (only for the second, third stage) or MSI test positive;
* Time interval to last chemotherapy is at least 1 month.
* 0-1 ECOG score
* The expected survival time is more than 4 months
* Peripheral blood cell culture showes the proliferation of lymphocytes

Exclusion Criteria:

* Participate in the plan or implementation of the research (including staff of HRYZ and the staff of the research center);
* Participate into other clinical studies at the same time, unless it is an observational (non - intervention) clinical study;
* Subjects may receive other systemic antitumor treatment during the study.
* Squamous or undifferentiated gastric cancer
* There were active bleeding, ulcers, gastrointestinal perforation, fistula, or arterial embolism in the gastrointestinal tract within 6 months.
* There were clinically significant gastrointestinal bleeding or venous thrombosis in three months before enrollment.
* End-stage cachexia patients;
* Patients with severe coagulation dysfunction;
* Patients with extensive abdominal adhesions;
* Patients with intestinal obstruction;
* Pregnancy or planned pregnancy;
* Refusing to provide blood specimens;
* Hypersensitivity to sodium citrate;
* Subjects have received allogeneic transplantation
* Subjects had clinical symptoms of central nervous system metastasis (such as brain edema, requiring hormone intervention, or progression of brain metastases)
* Subjects are using immunosuppressive agents, or whole body or absorbable local hormone therapy to achieve the aim of immunosuppression (dose >10mg/ days prednisone or other therapeutic hormones) and continue to use in the first 2 weeks before enrollment.
* Systemic or long-term application of immunomodulators, such as interferon, thymosin, and immunosuppressive drugs, in half a year.
* Subjects had been treated with MASCT or other cellular immunotherapy within a year.
* Subjects had any active autoimmune disease or a history of autoimmune disease.
* Active tuberculosis
* There is a big operation in 30 days before the first study treatment.
* Patients with active hepatitis B virus (HBV) infection (chronic or acute)
* The infection of active hepatitis C virus (HCV)
* Suffering from human immunodeficiency virus (HIV) or syphilis
* A history of peripheral nervous system disorder or a history of obvious mental disorders and central nervous system disorders
* Subjects had active infection or >38.5 degree of unexplained fever in the screening period and before the first administration.
* Chronic systemic diseases, such as liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease, or non controlled diabetes, hypertension, etc.
* There were other malignant tumors in 5 years, except for non melanin skin cancer and cervical carcinoma in situ
* There are heart symptoms or diseases that have not been well controlled.
* Subjects were known to have a history of psychotropic drug abuse, alcoholism, or drug abuse.
* According to the researchers, there are other factors that may lead to a halt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events（Safety） | The first 7 weeks
  All the local reactions, systemic reactions, adverse events and serious adverse events of all the patients obtained in 14 days after the first treatment cycle of the first course of treatment in this study

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu JI, Doctor, Principal Investigator — Cancer Hospital Affiliated to Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No